CLINICAL TRIAL: NCT01595165
Title: Effect of Subcostal Transversus Abdominis Plane Block on Early Postoperative Pain in Laparoscopic Cholecystectomy: Randomized, Controlled Trial
Brief Title: Transversus Abdominis Plane Block and Postoperative Pain After Laparoscopic Cholecystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Kim Sang-Hyun, Associate professor, Soonchunhyang University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: schbcanesthesia
Record Dates: First submitted 2012-05-07; First posted 2012-05-09 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-07

CONDITIONS: Laparoscopic Cholecystectomy; Postoperative Pain; Abdominal Muscles; Nerve Block
Keywords: laparoscopic cholecystectomy; ultrasound; transversus abdominis plane block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Placebo Comparator): Control group receiving saline instead of ropivacaine
  Interventions: Procedure: Placebo Ultrasound guided subcostal TAP block
- TAP (Experimental): TAP group receiving ropivacaine total of 150 mg at TAP under US
  Interventions: Procedure: Ultrasound guided subcostal TAP block

INTERVENTIONS:
Procedure: Ultrasound guided subcostal TAP block — Under ultrasound guidance0.375% ropivacaine 10 ml will be injected between rectus abdominis and transverse abdominis and same study solution will be injected at subcostal transversus abdominis plane. This block will be done bilaterally.
  Arms: TAP
Procedure: Placebo Ultrasound guided subcostal TAP block — Under ultrasound guidance saline 10 ml will be injected between rectus abdominis and transverse abdominis and same study solution will be injected at subcostal transversus abdominis plane. This block will be done bilaterally.
  Arms: Control

SUMMARY:
Transversus abdominis plane (TAP) block has gained popularity for the control of postoperative pain in various surgeries. Three studies showed inconsistent result on pain control after TAP block in laparoscopic cholecystectomy. The TAP technique used in these studies was classic ultrasound guided TAP block. Besides periumbilical incision, sub-xiphoid incision is usually made during laparoscopic cholecystectomy. As typical posterior TAP rarely extend above T8, the investigators undergo subcostal TAP block for this type of surgery. The investigators are going to investigate the effect of subcostal TAP on early postoperative pain after laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* Age 20-65 patients scheduled elective laparoscopic cholecystectomy

Exclusion Criteria:

* Patient refusal
* Allergy to ropivacaine
* Coagulopathy
* Morbid obesity (BMI>35 kg/m2)
* Previous abdominal surgery.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-07; Primary Completion 2012-12 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) 15 min after entering recovery room | 15 min after entering recovery room

SECONDARY OUTCOMES:
Fentanyl consumption at recovery room | Up to 3 hours until discharge from recovery room
Recovery room stay | Up to 3 hours from entering recovery room to discharge
Incidence of postoperative nausea and vomiting (PONV) | Up to 3 hours during recovery room stay
NRS at 4h, 24h, and 48 h after surgery | 4h, 24h, and 48 h after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Hyun Kim, M.D., Ph.D., Principal Investigator — Soonchunhyang University Hospital
Locations (1):
- Sang-Hyun Kim, Bucheon-si, Gyeonggi-do, South Korea